CLINICAL TRIAL: NCT00795184
Title: Detection Of Neoplastic Tissue in Barrett's Esophagus With In vivO Probe-based Confocal Endomicroscopy
Acronym: DONTBIOPCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mauna Kea Technologies (Industry)
Collaborators: Cellvizio Inc. (Industry); Emissary International LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: MKT-2008-BE-01
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Results first posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Barrett Syndrome; Barrett's Syndrome; Barrett's Esophagus; Barrett Esophagus; Adenocarcinoma
Keywords: Barrett's Esophagus; EsoGastroDuodenoscopy; Barrett's Carcinoma; adenocarcinoma; Cellvizio; endomicroscopy; random biopsy
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma | interventions — Diagnostic Imaging; Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Imaging Procedures HDWLE first NBI second and pCLE (Other): All patients undergo both endoscopic imaging procedures and then the endomicroscopy procedure; the endoscopic imaging procedures being performed back to back by two endoscopists, blinded to each other.
  Interventions: Device: Imaging procedures (NBI); Device: HDWLE; Device: pCLE
- Imaging Procedures NBI first HDWLE second and pCLE (Other): All patients undergo both endoscopic imaging procedures and then the endomicroscopy procedure; the endoscopic imaging procedures being performed back to back by two endoscopists, blinded to each other.
  Interventions: Device: Imaging procedures (NBI); Device: HDWLE; Device: pCLE

INTERVENTIONS:
Device: Imaging procedures (NBI) — Imaging procedures (pCLE) and (NBI) - All patients undergo both procedures back to back by two endoscopists, blinded to each other, in randomized order.
  Procedure 1: Standard endoscopic procedure The patient receives white light endoscopy (WLE) examination. All visible lesions are noted and photographed. No biopsy is taken until both procedures are complete.
  Procedure 2: NBI endoscopic procedure The patient receives a NBI endoscopy examination. All visible and NBI abnormal lesions are noted and photographed.
  After both procedures are complete and all sites are unblinded to both endoscopists. pCLE with Cellvizio and physical biopsies are performed at all sites plus 4 quadrant sites.
Device: HDWLE
Device: pCLE
  Other Names: Cellvizio

SUMMARY:
This study will collect data from patients routinely undergoing a endoscopic surveillance and Cellvizio endomicroscopy procedure due to confirmed Barrett's esophagus. The objective is to determine if endomicroscopy images collected using the marketed Cellvizio device may help endoscopists more accurately diagnose, in conjunction with traditional tissue sampling techniques, whether a suspected lesion is malignant or benign.

DETAILED DESCRIPTION:
This is a longitudinal observational study were imaging procedures are allocated in a random order to directly address the low sensitivity and specificity of enhanced macroscopic endoscopic imaging devices by determining whether probe-based Confocal Laser Endomicroscopy (pCLE), as a supplement to Narrow Band Imaging (NBI) can further improve sensitivity and specificity to a level that would be acceptable to avoid random biopsy, and better direct biopsy of suspicious areas. The study is also addressing pCLE as a supplement to standard white light endoscopy and random biopsy alone. In fact, the study is powered to evaluate per lesion sensitivity and specificity of confocal imaging as applied to lesions identified by white light endoscopy. Therefore, the study addresses the shortcomings of standard white light endoscopy (high number of random biopsies, less than ideal directed biopsy of suspicious areas) and the primary shortcomings of Narrow Band Imaging (NBI) (low specificity with resultant high false positives, again resulting in many unnecessary biopsies).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with documented or suspected Barrett's esophagus presenting for endoscopy
2. Age > 18 years
3. Ability to provide written, informed consent

Exclusion Criteria:

1. Presence of erosive esophagitis
2. Inability to obtain biopsies due to anticoagulation, varices, etc.
3. Allergy to fluorescein, pregnancy
4. Presence of an esophageal mass other than small 10mm or less nodules
5. Renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prateek Sharma, MD, Principal Investigator — Veterans Affairs Hospital, Kansas City
Locations (5):
- United States (3):
  - Mayo Clinic, Jacksonville, Florida
  - Veterans Affairs Hospital, Kansas City, Missouri
  - New York Presbyterian Hospital/Columbia University Medical Center, New York, New York
- Centre Hospitalier Universitaire, Nantes, France
- Klinikum rechts der Isar, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sharma P, Meining AR, Coron E, Lightdale CJ, Wolfsen HC, Bansal A, Bajbouj M, Galmiche JP, Abrams JA, Rastogi A, Gupta N, Michalek JE, Lauwers GY, Wallace MB. Real-time increased detection of neoplastic tissue in Barrett's esophagus with probe-based confocal laser endomicroscopy: final results of an international multicenter, prospective, randomized, controlled trial. Gastrointest Endosc. 2011 Sep;74(3):465-72. doi: 10.1016/j.gie.2011.04.004. Epub 2011 Jul 13. PMID 21741642

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | HDWLE First NBI Second and pCLE | NBI First HDWLE Second and pCLE
Started | 65 | 57
Completed | 57 (57 patients analysable, completed all 3 imaging procedures) | 44 (44 patients analysable, completed all 3 imaging procedures)
Not Completed | 8 | 13
Not completed — Tissue sampling incomplete/conclusive | 8 | 13

BASELINE CHARACTERISTICS:
Groups:
- Group 1: NBI-pCLE
Arm/Group | Group 1
Number analyzed (Participants) | 101
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.1 (11.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 87
Region of Enrollment [Number; unit: participants]
  France | 9
  United States | 62
  Germany | 30

OUTCOME MEASURES:

1. Primary Outcome: Comparative Histopathology-confirmed Measures of Per Lesion Sensitivity and Per Lesion Specificity, by Using pCLE Associated With WLE, or WLE Alone, for the Detection of High Grade Dysplasia and Early Carcinoma in Barrett's Esophagus.
Description: Comparative Histopathology-confirmed Measures of Per Lesion Sensitivity and Per Lesion Specificity, by Using Probe-based Confocal Laser Endomicroscopy (pCLE) Associated With White Light Endoscopy (WLE), or WLE Alone, for the Detection of High Grade Dysplasia and Early Carcinoma in Barrett's Esophagus.
Time Frame: Centralized histopathology confirmation within 4-6 weeks
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: Biopsy sites
Arm/Group | HDWLE | NBI (Narrow Band Imaging) | pCLE | HDWLE+NBI+pCLE | HDWLE+pCLE | HDWLE+NBI
Number analyzed (Participants) | 101 | 101 | 101 | 101 | 101 | 101
Number analyzed (Biopsy sites) | 874 | 874 | 874 | 874 | 874 | 874
percentage of lesions
  Sensitivity | 34.2 [25.7 to 42.7] | 41.7 [32.8 to 50.5] | 62.5 [53.8 to 71.2] | 75.8 [68.2 to 83.5] | 68.3 [60.0 to 76.7] | 45.0 [36.1 to 53.9]
  Specificity | 92.7 [90.8 to 94.6] | 90.5 [88.4 to 92.5] | 92.7 [90.8 to 94.6] | 84.2 [81.6 to 86.8] | 87.8 [85.5 to 90.1] | 88.2 [85.9 to 90.5]

ADVERSE EVENTS:
Time Frame: Acutely during the procedure - within the day
Groups:
- Group 1: NBI-pCLE or pCLE-NBI
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/122
Other Adverse Events (participants affected / at risk) | 0/122

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No